CLINICAL TRIAL: NCT05112523
Title: The Performance of Uroepithelial Cancer Risk Genes in the Necessity of Secondary Transurethral Resection of Bladder Tumor for High-risk Non-muscle-invasive Bladder Cancer: A Multicenter Clinical Trial
Brief Title: The Performance of Cancer Risk Genes in the Necessity of Secondary TURBT
Acronym: RE-TURBT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Hangzhou Jichenjunchuang Medical Laboratory Company (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2021-SR-277
Record Dates: First submitted 2021-10-07; First posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-10

CONDITIONS: Bladder Cancer
Keywords: Bladder Cancer; TURBT; Liquid biopsy; Uroepithelial cancer risk genes
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The genes of tumor exfoliated cells in urine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Investigators performed the Genetron Uro V1 test on the urine of patients before secondary TURBT and compared it with the final pathological results. To analyze the performance of the Genetron Uro V1 method in a study to predict the need for secondary TURBT in high-risk NMIBC patients and the correlation with patient's RFS and OS.

DETAILED DESCRIPTION:
The standard of treatment for patients with non-muscle invasive bladder cancer (NMIBC) is transurethral resection of bladder tumors (TURBT), with postoperative intravesical irrigation treatment options determined by the risk of recurrence. After TURBT surgery, tumor remnants are one of the most important causes of postoperative tumor recurrence. Studies have shown that secondary TURBT can detect residual bladder tumor lesions, obtain more accurate pathological staging, increase recurrence-free survival, improve patient prognosis, and enhance treatment outcomes. Current bladder cancer treatment guidelines recommend secondary TURBT for patients with (1) inadequate first TURBT (2) no muscle tissue in the first TURBT specimen, except for TaG1 and carcinoma in situ (3) stage T1 tumors (4) grade G3 tumors, except for carcinoma in situ. However, at present, the lack of screening methods for the population benefiting from secondary TURBT in clinical practice has led to some patients inevitably receiving overtreatment, increasing patient suffering, and financial costs, and raising the burden of government healthcare.

The genetic test for uroepithelial tumor risk (Genetron Uro V1) is a non-invasive liquid biopsy method based on urine samples, which has high diagnostic efficacy in patients with primary uroepithelial cancer. Investigators performed the Genetron Uro V1 test on the urine of patients before secondary TURBT and compared it with the final pathological results.

To analyze the performance of the Genetron Uro V1 method in a study to predict the need for secondary TURBT in high-risk NMIBC patients and the correlation with patient's RFS and OS.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a confirmed diagnosis of high-risk NMIBC at each study center:

   including (1) inadequate first TURBT; (2) absence of muscle tissue in the first TURBT specimen, except for TaG1 and carcinoma in situ alone; (3) stage T1 tumors; (4) grade G3 tumors, except for carcinoma in situ alone; (5) TaG1G2 meeting both multiple, recurrent, and >3 cm in diameter (or low-grade urothelial epithelial carcinoma)
2. gender is not limited.
3. age ≥ 18 years old.
4. the ability to provide a 100 ml standing urine sample within 3-6 weeks after the first TURBT and before the secondary transurethral resection.
5. agree to provide basic personal clinical information and pathological and imaging data for use in scientific research and sign an informed consent form related to scientific research.
6. consent to perform the genetic testing services involved in the trial.
7. agree to provide monitoring results in the follow-up relapse monitoring process.

Exclusion Criteria:

1. patients with other non-uroepithelial malignancies (including prostate cancer and renal cell carcinoma).
2. patients who failed to undergo secondary transurethral resection.
3. patients with incomplete information on sample pathology.
4. patients with contaminated samples.
5. Patients whose urine samples fail quality control and cannot be re-sampled for valid reasons.
6. Patients whose samples cannot complete the test due to reasonable cause.
7. any condition that, in the opinion of the investigator, may harm the subject or cause the subject to be unable to meet or perform the requirements of the study.
8. Patients who are unable to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receive a confirmed diagnosis of high-risk NMIBC at each study center and undergo the first TURBT
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-12-20 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Concordance analysis of Genetron Uro V1 assay results with gold standard results of secondary TURBT histopathology | Through study completion, an average of 1 year
  Through Concordance analysis of Genetron Uro V1 assay results with gold standard results of secondary TURBT histopathology, the sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV) of Genetron Uro V1 detected before secondary TURBT are measured.

SECONDARY OUTCOMES:
Overall survival | 2 years after surgery
  To analyze the performance of the Genetron Uro V1 method in a study to predict the correlation with patient OS.
Recurrence-free survival | 2 years after surgery
  To analyze the performance of the Genetron Uro V1 method in a study to predict the correlation with patient RFS.

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Lv, MD，PHD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The first affiliated hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No